CLINICAL TRIAL: NCT05078632
Title: Montreal Toulouse 86 Test Modified to be Used With Eye Tracking: Test Automation and Eye Course in Healthy Volunteers and Intensive Care Patients
Brief Title: Montreal Toulouse Test With Eye Tracking in Intensive Care Unit to Evaluate Comprehension
Acronym: MEXICO
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR190027-MEXICO
Record Dates: First submitted 2021-06-23; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Critical Care
Keywords: eye tracking; critical care; comprehension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: healthy volunteers
  Interventions: Other: Montreal-Toulouse Test adapted in eye tracking
- intensive care patient: patient hospitalized in intensive care unit
  Interventions: Other: Montreal-Toulouse Test adapted in eye tracking

INTERVENTIONS:
Other: Montreal-Toulouse Test adapted in eye tracking — participant pass an eye tracking test to evaluate comprehension

SUMMARY:
Assessment of the level of oral comprehension of the intensive care patient is essential to improve their care because they have often troubles like delirium.

DETAILED DESCRIPTION:
Assessment of the level of oral comprehension of the intensive care patient is essential to improve their care because they have often troubles like delirium.

ELIGIBILITY:
Inclusion Criteria:

* French speaker, RASS (Richmond Agitation-sedation scale) between -1 and +1, agree for participation

Exclusion Criteria:

* neurovisual disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and patient hospitalized in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Establish eye tracking standards for the test | during hospitalization in intensive care
  fixation time measurement in the defined area of interest

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia BODET-CONTENTIN, MD-PhD, Principal Investigator — University Hospital of TOURS
Locations (1):
- CHU Tours, Tours, France